CLINICAL TRIAL: NCT03453554
Title: Evaluating a Digital Memory Notebook Intervention to Improve Independence and Quality of Life
Brief Title: Evaluating a Digital Memory Notebook App to Improve Functional Independence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Washington State University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AZ150096
Record Dates: First submitted 2018-02-07; First posted 2018-03-05 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-02

CONDITIONS: Mild Cognitive Impairment
Keywords: technology; activities of daily living; everyday functioning; quality of life; memory impairment
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DMN/Smart Home Partnership (Experimental): Participants will learn how to use a digital memory notebook partnered with smart environment prompting technology to support everyday activities of daily living and reduce problems associated with memory deficits.
  Interventions: Other: Digital Notebook app; Other: Smart Home Prompting
- Digital Memory Notebook app (Active Comparator): Participants will learn how to use a Digital Memory Notebook app to support everyday activities of daily living and reduce problems associated with memory deficits.
  Interventions: Other: Digital Notebook app

INTERVENTIONS:
Other: Digital Notebook app — Training in use of Digital Memory Notebook app
Other: Smart Home Prompting — Smart-home sensor based activity-aware prompting to support digital memory notebook app use
  Arms: DMN/Smart Home Partnership

SUMMARY:
This study will investigate the efficacy of a smart home / digital memory notebook (DMN) partnership that will allow for real-time intervention and thereby facilitate acquisition and use of the DMN to support everyday independence. The DMN is an app that is installed on a mobile tablet. The smart home technology discovers and recognizes generalizable activities and provides information about functional status and health-related variables for older adult participants. This study will examine how smart home prompts affect individuals' DMN use, ability to maintain activity routines, and overall wellbeing. Prompts will center on helping users organize and schedule daily activities, record both routine and uncommon events that may need to be remembered, and record activities performed and important associated event information (e.g., when, what, where). Prompting will help to promote everyday functional independence by encouraging frequent and regular notebook use and reducing memory difficulties. The DMN will also help to support functional independence by notifying individuals about appointments or prompting individuals to initiate important activities of daily living (e.g., take medications).

This study will also involve a machine learning technique to gain a better understanding of the contexts in which individuals adhere or do not adhere to the prompts. This activity-aware intervention will be deployed in the homes of older adults with memory difficulties, to assess the usability of the technology as well as to evaluate in a naturalistic setting the efficacy of the technology for increasing everyday functional independence and quality of life and decreasing care-partner burden. This contribution is significant because it will demonstrate that intelligent technologies can improve the efficacy of traditional memory rehabilitation techniques, extend functional independence, reduce caregiver burden, and improve quality of life.

DETAILED DESCRIPTION:
Approximately 30 older adults who complain of memory problems will be recruited for this study. Over the course of six months, participants will complete questionnaires, open-ended questions, and cognitive and motor screens. Participants will also undergo training to learn to use a DMN to support daily activities and will continue to use the DMN for three months following training. Additionally, half of the participants' homes will be equipped with our "smart home in a box" technology that will support DMN use with context-aware prompting technology.

During month one, participants in both conditions will complete a cognitive and motor screen as well as questionnaires assessing depression, quality of life, coping, everyday memory, and functional abilities. Care-partners/informants (when available) will also complete the same questionnaires as well as an additional questionnaire about caregiver burden. The questionnaires will be administered monthly (6x total) for the duration of the study.

During month two, graduate students will train study participants to use the DMN using a training manual and workbook in 6-8 training sessions (depending on participants comfort with the DMN) over 3-4 weeks. Supervision will include review of audiotapes and use of a checklist to monitor fidelity of the training content and process. Participants and care-partners will also answer open-ended questions designed to help improve the DMN and its training procedure as well as the prompting technology and its integration with the DMN at each assessment period. In addition, participants and care-partners will complete questionnaires about their satisfaction and perception of ease of use of the DMN and interface as well as a questionnaire concerning likeability and cognitive demand.

During months three through five, data collection will continue. Participants in the smart home condition will use the DMN in conjunction with prompting technology for the third month, only the DMN for the fourth month, and again the DMN and prompting technology for the fifth month. Control participants will use only the DMN for all three months. Control participants will rely on traditional methods (e.g., time-based alarm cues, sticky notes) to support DMN use rather than activity-aware prompting technology.

During month six, participants will complete a post-test cognitive and motor screen identical to the initial screen. Participants will also complete the set of the previously described questionnaires and open-ended questions.

ELIGIBILITY:
Inclusion Criteria:

* age 40+
* memory problems documented by self-report
* memory problems documented by cognitive data (i.e., memory testing > 1 std below expectations for age and education)
* English speaking

Exclusion Criteria:

* unable to provide own informed consent
* lack insight/awareness that are experiencing memory difficulties

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Digital Memory Notebook Use | Change will be assessed between monthly time points (1-, 2-, 3-, 4-, and 5-months).
  Mean number of monthly DMN entries made and mean number of monthly DMN uses as measured continuously via the DMN app will be totaled to form a monthly DMN Memory Notebook use score.
Quality of Life | Total change in quality of life as measured by QOL-AD (range 13 [poor]-52 [best]) between baseline and monthly time points (1-, 2-, 3-, 4-, and 5-months).
  The Quality of Life-Alzheimer's disease (QOL-AD; Logsdon, 1996) scale will be used to measure quality of life and subjective well-being.
Activities of Daily Living | Total change in functional status as measured by IADL-C (range 27 [best]-216 [poor]) between baseline and monthly time points (1-, 2-, 3-, 4-, and 5-months).
  The Instrumental Activities of Daily Living- Compensation (IADL-C; Schmitter-Edgecombe, Parsey, & Lamb, 2014) will be used to provide an estimate of functional difficulties.
Caregiver Burden | Total change in caregiver burden as measured by CBS (range 0 [best]-96 [poor]) between baseline and monthly time points (1-, 2-, 3-, 4-, and 5-months).
  The Caregiver Burden Scale (CBS; Elmstahl et al., 1996) will be used to assess caregiver burden experienced by participants' care-partners.

SECONDARY OUTCOMES:
Coping self-efficacy | Total change in coping self-efficacy as measured by CSES (range 0 [poor]-130 [best]) between baseline and monthly time points (1-, 2-, 3-, 4-, and 5-months)
  The Coping Self Efficacy Scale (CSES) assesses participants' perceived abilities to cope with life challenges.
Cognitive functioning | Total change in cognitive functioning as measured by RBANS (total score) at baseline and end of intervention (6 Months)
  Neuropsychological assessment: Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Schmitter-Edgecombe, PhD, Principal Investigator — Washington State University
Locations (1):
- Washington State University - Pullman, Pullman, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luna C, Cook DJ, Schmitter-Edgecombe M. But will they use it? Predictors of adoption of an electronic memory aid in individuals with amnestic mild cognitive impairment. Neuropsychology. 2023 Nov;37(8):955-965. doi: 10.1037/neu0000898. Epub 2023 Mar 20. PMID 36939601
- [Derived] Schmitter-Edgecombe M, Brown K, Luna C, Chilton R, Sumida CA, Holder L, Cook D. Partnering a Compensatory Application with Activity-Aware Prompting to Improve Use in Individuals with Amnestic Mild Cognitive Impairment: A Randomized Controlled Pilot Clinical Trial. J Alzheimers Dis. 2022;85(1):73-90. doi: 10.3233/JAD-215022. PMID 34776442
- [Derived] Chudoba LA, Church AS, Dahmen JB, Brown KD, Schmitter-Edgecombe M. The development of a manual-based digital memory notebook intervention with case study illustrations. Neuropsychol Rehabil. 2020 Oct;30(9):1829-1851. doi: 10.1080/09602011.2019.1611606. Epub 2019 May 3. PMID 31046586